CLINICAL TRIAL: NCT01411527
Title: The COPENHAGEN Puberty Study Providing Normative Data of Healthy Danish Children and Adolescents
Brief Title: The COPENHAGEN Puberty Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); European Commission (Other)
Responsible Party: Principal Investigator, Anders Juul, Professor, Rigshospitalet, Denmark
Other Study IDs: KF01282214
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Puberty
Keywords: Hormones; Endocrine Disrupters; Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, white cells, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross- sectional cohort: Schools were randomly selected and 6203 children (50.0 % girls) were invited to participate. 1864 (1097 girls and 767 boys) (age 5.6-20.0 years) were included, resulting in an overall participation-rate of 30%. Blood samples were drawn, and a thorough clinical examination was performed in all participating children
- Longitudinal cohort: 209 healthy Danish children (108 girls), were examined and blood samples were drawn every 6 months. In july 2011, the mean (range) number of examinations per child was 7 (2-10).
  116 (63 boys and 53 girls) continued from the cross sectional study to the longitudinal study. Thus, the total number of participants in The COPENHAGEN Puberty Study was 2020 children.

SUMMARY:
By clinical examinations and withdrawing of blood samples from a large number of healthy Danish children, this study will reveal if age of pubertal onset is declining. Furthermore, the extensive normative data will provide detailed insight into normal ranges and individual changes of anthropometrics and hormone levels in healthy children during childhood and adolescence.

DETAILED DESCRIPTION:
The COPENHAGEN Puberty Study is a combined cross sectional and longitudinal study of healthy Danish children.

All children will be thoroughly examined and blood- and urine samples will be collected at every visit. The families fill out questionaires.

Physical examination: Height; sitting-height; weight; circumference of waist, hip, arm; measurement of fatfolds (biceps, triceps, flank, subscapularis); voice-break (yes/no), blood pressure; pubertal staging according to Tanners classification: breast development (B1-B5), genitalia development boys (G1-G5), pubic hair development (PH1-PH5), axillary hair (yes/no), sweat (yes/no), acne (yes/no

Urine sample: For measurement of FSH, LH and endocrine disrupters.

Blood sample: For measurement of hormone levels (FSH, LH, estradiol, SHBG, testosterone, DHEAS, androstenedione, inhibin A, inhibin B, Insl3, kisspeptin, ghrelin, leptin, IGF-1, IGFBP3, TSH, T4, Free T4, T3, HbA1C, calcium-ion, PTH, phosphate, 25-OH-vitamine D, AMH), endocrine disrupters (PCB´s, dioxines, parabens, phthalates), isolation of DNA and RNA to evaluate relevant polymorphisms.

Questionaire: regarding information of previous growth and health.

ELIGIBILITY:
Inclusion Criteria:

* all children accepting to participate were included

Exclusion Criteria:

* no children were excluded from examination or blood sampling. In case of chronic diseases, medical treatment, or ethnicity the children may be excluded from specific final data analysis.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In the cross sectional study, all children at randomly selected schools in Copenhagen were invited (6203 children). 1864 accepted to participate.
  In the longitudinal study, children at two schools with the highest participating rate were invited to participate in the follow-up study. Ongoing recruitment was continued until at least 100 boys and 100 girls were enrolled in the logitudinal study.
Sampling Method: Non-Probability Sample
Enrollment: 1957 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, PhD, DMSc, Study Director — Rigshospitalet, dept. of Growth and Reproduction
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Courant F, Aksglaede L, Antignac JP, Monteau F, Sorensen K, Andersson AM, Skakkebaek NE, Juul A, Bizec BL. Assessment of circulating sex steroid levels in prepubertal and pubertal boys and girls by a novel ultrasensitive gas chromatography-tandem mass spectrometry method. J Clin Endocrinol Metab. 2010 Jan;95(1):82-92. doi: 10.1210/jc.2009-1140. Epub 2009 Nov 20. PMID 19933393
- [Result] Aksglaede L, Sorensen K, Petersen JH, Skakkebaek NE, Juul A. Recent decline in age at breast development: the Copenhagen Puberty Study. Pediatrics. 2009 May;123(5):e932-9. doi: 10.1542/peds.2008-2491. PMID 19403485
- [Result] Sorensen K, Aksglaede L, Petersen JH, Juul A. Recent changes in pubertal timing in healthy Danish boys: associations with body mass index. J Clin Endocrinol Metab. 2010 Jan;95(1):263-70. doi: 10.1210/jc.2009-1478. Epub 2009 Nov 19. PMID 19926714
- [Result] Sorensen K, Aksglaede L, Munch-Andersen T, Aachmann-Andersen NJ, Petersen JH, Hilsted L, Helge JW, Juul A. Sex hormone-binding globulin levels predict insulin sensitivity, disposition index, and cardiovascular risk during puberty. Diabetes Care. 2009 May;32(5):909-14. doi: 10.2337/dc08-1618. Epub 2009 Feb 5. PMID 19196890
- [Result] Juul A, Sorensen K, Aksglaede L, Garn I, Rajpert-De Meyts E, Hullstein I, Hemmersbach P, Ottesen AM. A common deletion in the uridine diphosphate glucuronyltransferase (UGT) 2B17 gene is a strong determinant of androgen excretion in healthy pubertal boys. J Clin Endocrinol Metab. 2009 Mar;94(3):1005-11. doi: 10.1210/jc.2008-1984. Epub 2008 Dec 16. PMID 19088161
- [Result] Sorensen K, Aksglaede L, Munch-Andersen T, Aachmann-Andersen NJ, Leffers H, Helge JW, Hilsted L, Juul A. Impact of the growth hormone receptor exon 3 deletion gene polymorphism on glucose metabolism, lipids, and insulin-like growth factor-I levels during puberty. J Clin Endocrinol Metab. 2009 Aug;94(8):2966-9. doi: 10.1210/jc.2009-0313. Epub 2009 May 5. PMID 19417039
- [Result] Sorensen K, Aksglaede L, Petersen JH, Leffers H, Juul A. The exon 3 deleted growth hormone receptor gene is associated with small birth size and early pubertal onset in healthy boys. J Clin Endocrinol Metab. 2010 Jun;95(6):2819-26. doi: 10.1210/jc.2009-2484. Epub 2010 Apr 9. PMID 20382688
- [Result] Sorensen K, Mouritsen A, Mogensen SS, Aksglaede L, Juul A. Insulin sensitivity and lipid profiles in girls with central precocious puberty before and during gonadal suppression. J Clin Endocrinol Metab. 2010 Aug;95(8):3736-44. doi: 10.1210/jc.2010-0731. Epub 2010 May 19. PMID 20484471
- [Result] Hagen CP, Aksglaede L, Sorensen K, Main KM, Boas M, Cleemann L, Holm K, Gravholt CH, Andersson AM, Pedersen AT, Petersen JH, Linneberg A, Kjaergaard S, Juul A. Serum levels of anti-Mullerian hormone as a marker of ovarian function in 926 healthy females from birth to adulthood and in 172 Turner syndrome patients. J Clin Endocrinol Metab. 2010 Nov;95(11):5003-10. doi: 10.1210/jc.2010-0930. Epub 2010 Aug 18. PMID 20719830
- [Result] Aksglaede L, Sorensen K, Boas M, Mouritsen A, Hagen CP, Jensen RB, Petersen JH, Linneberg A, Andersson AM, Main KM, Skakkebaek NE, Juul A. Changes in anti-Mullerian hormone (AMH) throughout the life span: a population-based study of 1027 healthy males from birth (cord blood) to the age of 69 years. J Clin Endocrinol Metab. 2010 Dec;95(12):5357-64. doi: 10.1210/jc.2010-1207. Epub 2010 Sep 15. PMID 20843948
- [Result] Mogensen SS, Aksglaede L, Mouritsen A, Sorensen K, Main KM, Gideon P, Juul A. Diagnostic work-up of 449 consecutive girls who were referred to be evaluated for precocious puberty. J Clin Endocrinol Metab. 2011 May;96(5):1393-401. doi: 10.1210/jc.2010-2745. Epub 2011 Feb 23. PMID 21346077
- [Result] Aksglaede L, Christiansen P, Sorensen K, Boas M, Linneberg A, Main KM, Andersson AM, Skakkebaek NE, Juul A. Serum concentrations of Anti-Mullerian Hormone (AMH) in 95 patients with Klinefelter syndrome with or without cryptorchidism. Acta Paediatr. 2011 Jun;100(6):839-45. doi: 10.1111/j.1651-2227.2011.02148.x. Epub 2011 Feb 25. PMID 21251056
- [Result] Frederiksen H, Aksglaede L, Sorensen K, Nielsen O, Main KM, Skakkebaek NE, Juul A, Andersson AM. Bisphenol A and other phenols in urine from Danish children and adolescents analyzed by isotope diluted TurboFlow-LC-MS/MS. Int J Hyg Environ Health. 2013 Nov;216(6):710-20. doi: 10.1016/j.ijheh.2013.01.007. Epub 2013 Mar 13. PMID 23491025
- [Result] Mouritsen A, Hagen CP, Sorensen K, Aksglaede L, Mieritz MG, Main KM, Almstrup K, Rajpert-De Meyts E, Juul A. Androgen receptor CAG repeat length is associated with body fat and serum SHBG in boys: a prospective cohort study. J Clin Endocrinol Metab. 2013 Mar;98(3):E605-9. doi: 10.1210/jc.2012-3778. Epub 2013 Feb 7. PMID 23393169
- [Result] Mouritsen A, Aksglaede L, Soerensen K, Hagen CP, Petersen JH, Main KM, Juul A. The pubertal transition in 179 healthy Danish children: associations between pubarche, adrenarche, gonadarche, and body composition. Eur J Endocrinol. 2012 Dec 31;168(2):129-36. doi: 10.1530/EJE-12-0191. Print 2013 Feb. PMID 23093700
- [Result] Hilsted L, Rustad P, Aksglaede L, Sorensen K, Juul A. Recommended Nordic paediatric reference intervals for 21 common biochemical properties. Scand J Clin Lab Invest. 2013 Feb;73(1):1-9. doi: 10.3109/00365513.2012.721519. Epub 2012 Sep 26. PMID 23013046
- [Result] Mieritz MG, Frederiksen H, Sorensen K, Aksglaede L, Mouritsen A, Hagen CP, Skakkebaek NE, Andersson AM, Juul A. Urinary phthalate excretion in 555 healthy Danish boys with and without pubertal gynaecomastia. Int J Androl. 2012 Jun;35(3):227-35. doi: 10.1111/j.1365-2605.2012.01279.x. PMID 22612475
- [Result] Frederiksen H, Sorensen K, Mouritsen A, Aksglaede L, Hagen CP, Petersen JH, Skakkebaek NE, Andersson AM, Juul A. High urinary phthalate concentration associated with delayed pubarche in girls. Int J Androl. 2012 Jun;35(3):216-26. doi: 10.1111/j.1365-2605.2012.01260.x. Epub 2012 Mar 19. PMID 22428786
- [Result] Hagen CP, Aksglaede L, Sorensen K, Mouritsen A, Andersson AM, Petersen JH, Main KM, Juul A. Individual serum levels of anti-Mullerian hormone in healthy girls persist through childhood and adolescence: a longitudinal cohort study. Hum Reprod. 2012 Mar;27(3):861-6. doi: 10.1093/humrep/der435. Epub 2012 Jan 2. PMID 22215627
- [Result] Busch AS, Hagen CP, Main KM, Pereira A, Corvalan C, Almstrup K, Mericq V, Juul A. Genetic Variation of Follicle-Stimulating Hormone Action Is Associated With Age at Testicular Growth in Boys. J Clin Endocrinol Metab. 2017 May 1;102(5):1740-1749. doi: 10.1210/jc.2016-4013. PMID 28323923
- [Result] Busch AS, Hagen CP, Almstrup K, Juul A. Circulating MKRN3 Levels Decline During Puberty in Healthy Boys. J Clin Endocrinol Metab. 2016 Jun;101(6):2588-93. doi: 10.1210/jc.2016-1488. Epub 2016 Apr 8. PMID 27057785
- [Result] Almstrup K, Lindhardt Johansen M, Busch AS, Hagen CP, Nielsen JE, Petersen JH, Juul A. Pubertal development in healthy children is mirrored by DNA methylation patterns in peripheral blood. Sci Rep. 2016 Jun 28;6:28657. doi: 10.1038/srep28657. PMID 27349168
- [Derived] Busch AS, Ljubicic ML, Upners EN, Fischer MB, Hagen CP, Fluck CE, Johannsen TH, Frederiksen H, Juul A. Serum steroid metabolome dynamics in infancy: a longitudinal cohort study of healthy infants. Eur J Endocrinol. 2025 Sep 30;193(4):403-411. doi: 10.1093/ejendo/lvaf193. PMID 40974100
- [Derived] Sorensen K, Hagen CP, Juul A. Higher peak height velocity in early maturing girls depends on insulin rather than fat mass or IGF-I. Eur J Endocrinol. 2024 Sep 30;191(4):381-388. doi: 10.1093/ejendo/lvae115. PMID 39292994
- [Derived] Busch AS, Ljubicic ML, Upners EN, Fischer MB, Kolby N, Eckert-Lind C, Jespersen K, Andersson AM, Frederiksen H, Johannsen TH, Hegaard HK, Sharif H, Hagen CP, Juul A. Cohort profile: The COPENHAGEN Minipuberty Study-A longitudinal prospective cohort of healthy full-term infants and their parents. Paediatr Perinat Epidemiol. 2021 Sep;35(5):601-611. doi: 10.1111/ppe.12777. Epub 2021 Jun 22. PMID 34156716
- [Derived] Albrethsen J, Ljubicic ML, Juul A. Longitudinal Increases in Serum Insulin-like Factor 3 and Testosterone Determined by LC-MS/MS in Pubertal Danish Boys. J Clin Endocrinol Metab. 2020 Oct 1;105(10):dgaa496. doi: 10.1210/clinem/dgaa496. PMID 32761207
- [Derived] Busch AS, Hojgaard B, Hagen CP, Teilmann G. Obesity Is Associated with Earlier Pubertal Onset in Boys. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz222. doi: 10.1210/clinem/dgz222. PMID 31761939
- [Derived] Busch AS, Hollis B, Day FR, Sorensen K, Aksglaede L, Perry JRB, Ong KK, Juul A, Hagen CP. Voice break in boys-temporal relations with other pubertal milestones and likely causal effects of BMI. Hum Reprod. 2019 Aug 1;34(8):1514-1522. doi: 10.1093/humrep/dez118. PMID 31348498
- [Derived] Busch AS, Hagen CP, Assens M, Main KM, Almstrup K, Juul A. Differential Impact of Genetic Loci on Age at Thelarche and Menarche in Healthy Girls. J Clin Endocrinol Metab. 2018 Jan 1;103(1):228-234. doi: 10.1210/jc.2017-01860. PMID 29077908
- [Derived] Kolby N, Busch AS, Aksglaede L, Sorensen K, Petersen JH, Andersson AM, Juul A. Nocturnal Urinary Excretion of FSH and LH in Children and Adolescents With Normal and Early Puberty. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3830-3838. doi: 10.1210/jc.2017-01192. PMID 28938419
- [Derived] Lindhardt Johansen M, Hagen CP, Mieritz MG, Wolthers OD, Heuck C, Petersen JH, Juul A. Pubertal Progression and Reproductive Hormones in Healthy Girls With Transient Thelarche. J Clin Endocrinol Metab. 2017 Mar 1;102(3):1001-1008. doi: 10.1210/jc.2016-2871. PMID 28009526
- [Derived] Bisgaard A, Sorensen K, Johannsen TH, Helge JW, Andersson AM, Juul A. Significant gender difference in serum levels of fibroblast growth factor 21 in Danish children and adolescents. Int J Pediatr Endocrinol. 2014;2014(1):7. doi: 10.1186/1687-9856-2014-7. Epub 2014 May 23. PMID 24883065
- [Derived] Nielsen J, Jensen RB, Juul A. Increased sex hormone-binding globulin levels in children and adolescents with thyrotoxicosis. Horm Res Paediatr. 2013;79:157-61. doi: 10.1159/000348837. Epub 2013 Mar 27. PMID 23548728
- [Derived] Hagen CP, Sorensen K, Anderson RA, Juul A. Serum levels of antimullerian hormone in early maturing girls before, during, and after suppression with GnRH agonist. Fertil Steril. 2012 Nov;98(5):1326-30. doi: 10.1016/j.fertnstert.2012.07.1118. Epub 2012 Aug 14. PMID 22901847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-sectional study: All pupils at 10 different schools in the Copenhagen area were invited to participate.
  Longitudinal study: All pupils from 2 of the 10 schools were invited to participate in the follow up study. This includes pupils that have been recruited to the cross-sectional part. (see footnote)
Pre-assignment Details: No participants were excluded
Groups:
- Cross- Sectional Cohort: Schools were randomly selected. Blood samples were drawn, and a thorough clinical examination was performed in all participating children
- Longitudinal Cohort: Healthy Danish children were examined and blood samples were drawn every 6 months.
Period: Overall Study
Arm/Group | Cross- Sectional Cohort | Longitudinal Cohort
Started | 1864 | 93
Completed (116 participants were later transferred to the longitudinal cohort) | 1864 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Longitudinal Cohort: 209 healthy Danish children (108 girls), were examined and blood samples were drawn every 6 months. In july 2011, the mean (range) number of examinations per child was 7 (2-10).
  116 (63 boys and 53 girls) continued from the cross sectional study to the longitudinal study.
- Total: Total of all reporting groups
Arm/Group | Cross- Sectional Cohort | Longitudinal Cohort | Total
Number analyzed (Participants) | 1748 | 209 | 1957
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1748 | 209 | 1957
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.8 [5.6 to 20] | 11.8 [5.6 to 20] | 11.8 [5.6 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1044 | 108 | 1152
  Male | 704 | 101 | 805
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1748 | 209 | 1957
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 1748 | 209 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pubertal Onset
Description: Pubertal onset (according to Tanner stageing - Marshall & Tanner 1969 and 1970), i.e. Tanner stages B2+ or G2+ [Tanner stages included genital stages 1-5 as well as pubic hairs tages 1-6]
  Data of both arms were pooled for calculation of means.
Time Frame: up to 8 year period.
Population: Population
Measure: Mean (95% Confidence Interval); unit: years
Groups:
- Cross- Sectional Cohort: Schools were randomly selected and 6203 children (50.0 % girls) were invited to participate (overall participation-rate: 30%). Blood samples were drawn, and a thorough clinical examination was performed in all participating children
- Longitudinal Cohort: 209 healthy Danish children (108 girls), were examined and blood samples were drawn every 6 months.
Arm/Group | Cross- Sectional Cohort | Longitudinal Cohort
Number analyzed (Participants) | 1748 | 209
years
  Girls | 9.86 [9.70 to 10.01] | 9.86 [9.70 to 10.01]
  Boys | 11.66 [11.49 to 11.82] | 11.66 [11.49 to 11.82]

ADVERSE EVENTS:
Time Frame: 6 years
Description: No serious and/or other adverse events did occur
Groups:
- Population: This is a descriptive study elucidating normal variation. Therefore, the study population is not grouped
Arm/Group | Population
All-Cause Mortality (participants affected / at risk) | 0/1957
Serious Adverse Events (participants affected / at risk) | 0/1957
Other Adverse Events (participants affected / at risk) | 0/1957

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No